CLINICAL TRIAL: NCT00791492
Title: An Open-Label Extension Of Study Fx-005 Evaluating Long-Term Safety And Clinical Outcomes Of Fx-1006A In Patients With Transthyretin Amyloid Polyneuropathy
Brief Title: An Extension of Study Fx-005 Evaluating Long-Term Safety And Clinical Outcomes Of Fx-1006A In Patients With Transthyretin Amyloid Polyneuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX-006; B3461021
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Familial Amyloid Polyneuropathy; ATTR-PN
Keywords: FAP; Familial Amyloid Polyneuropathy; ATTR-PN; transthyretin; TTR; amyloid; polyneuropathy; familial; hereditary; amyloidosis; FoldRx
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Alzheimer Disease; Polyneuropathies; Amyloidosis | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fx-1006A (Experimental)
  Interventions: Drug: Fx-1006A

INTERVENTIONS:
Drug: Fx-1006A — Fx-1006A 20mg soft gelatin capsule administered orally once daily (at the same time each day) for 12 months.

SUMMARY:
This study is designed to determine the long-term safety and tolerability of Fx-1006A as well as the effects of Fx-1006A on clinical outcomes in patients with ATTR-PN.

All patients who enroll in this extension study will receive once-daily oral 20 mg Fx-1006A for 12 months; therefore, patients randomized to placebo in Study Fx-005 will cross over to active drug (Fx-1006A 20 mg) during this study. However, patients and their families as well as clinical Investigators and their clinical site staff will remain blinded to the original Fx-005 treatment assignment. It is intended that there will be no interruption in study medication administration between the two studies. The majority of safety and clinical outcomes assessments will be identical to those evaluated in Study Fx-005. Additional assessments for this open-label extension study include 24-hour Holter monitoring and skin biopsy for IENF; patients will be required to provide written informed consent to participate in this open-label extension study prior to having these additional procedures performed.

The values obtained from procedures and evaluations conducted during the Month 18 visit of Study Fx-005 will be used as the Baseline values for this open-label extension study. The Baseline assessments of IENF and Holter monitoring may be conducted at either day of the Month 18 visit days of Study Fx-005, but prior to the first Fx-1006A dose in this open-label extension study. Clinic Visits will be conducted at Week 6 (± 2 days), and Month 3 (± 1 week), Month 6 (± 2 weeks), and Month 12 (± 2 weeks). Monthly telephone contacts (± 1 week of the scheduled date) will be made during months in which no investigative site visits are scheduled (Months 2, 4, 5, 7, 8, 9, 10, and 11) for assessment of adverse events and concomitant medications.

Neurological evaluation by NIS-LL will be performed at Months 6 and 12. The NIS-LL will be assessed by utilizing the average of two successive NIS-LL clinical assessment scores obtained at least 24 hours apart within a one week period for each study visit. A dedicated neurologist will be required to perform NIS-LL scoring across all time-points for each individual patient enrolled in the study.

Quality of life utilizing the Norfolk QOL-DN will be assessed at Months 6 and 12 (based on the total score as well as the five individual domains of the questionnaire).

QST (utilizing CASE IV), NCS, HRDB, mBMI, and echocardiography will be conducted at Months 6 and 12. Holter monitoring will be conducted at Baseline and Months 6 and 12. Biopsies for IENF will be obtained at Baseline only. Assessments of troponin I and NT-pro-BNP levels will be made at each study visit.

Blood samples for pharmacokinetic assessments (Fx-1006A concentrations as well as calculated steady-state parameters) and pharmacodynamic assessments (TTR stabilization) will be collected at Week 6 and Months 6 and 12.

Safety and tolerability will be assessed throughout the study. Vital signs, 12-lead ECG, blood and urine samples for clinical laboratory tests (serum chemistry, hematology, coagulation panel, urinalysis, and urine pregnancy testing), adverse events, and concomitant medications will be assessed at each study visit. Eye examinations (including fundal photography) will be conducted at Months 6 and 12. Abbreviated physical examinations will be conducted at Week 6, and Months 3 and 6, and a complete physical examination will be conducted at Month 12.

All patients will be contacted by telephone 30 days (± 1 week) after the last dose of study medication for assessment of adverse events and concomitant medications.

Patients who complete the Month 12 visit of this open-label study may be allowed to continue receiving Fx-1006A under a compassionate use program.

Patients who discontinue from the study at any time after enrollment (i.e., early termination) will have final safety assessments performed at the time of discontinuation. Any patient discontinuing after the Month 6 visit will have all safety and clinical outcomes assessments scheduled for the Month 12 visit performed.

ELIGIBILITY:
Inclusion Criteria:

Male and non-pregnant female patients meeting all of the following criteria are eligible for enrollment in this study:

* Patient has completed the Month 18 visit of Study Fx-005.
* If female, patient is post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide) throughout the study. (A condom alone is not considered an acceptable method of birth control.) If male with a female partner of childbearing potential, willing to use an acceptable method of birth control for the duration of the study. For both females and males, acceptable birth control must be used for at least 3 months after the last dose of study medication.
* Patient is, in the opinion of the investigator, willing and able to comply with the study medication regimen and all other study requirements.
* Patient agrees not to participate in another investigational drug or device study while participating in this open-label extension study.

Exclusion Criteria:

Patients meeting any of the exclusion criteria will not be enrolled in the study:

* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs), defined as greater than 3-4 times/month (ibuprofen and nimesulide will be permitted).
* If female, patient is pregnant or breast feeding.
* Patient has liver function test abnormalities: alanine transaminases (ALT) and/or aspartate transaminases (AST) >2 times upper limit of normal (ULN) that in the medical judgment of the investigator are due to reduced liver function or active liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Packman, Study Director — FoldRx Pharmaceuticals, Inc.
Locations (11):
- Argentina (2):
  - FLENI Departamento de Hepatología y Transplante de Organos, Buenos Aires
  - FLENI-Hepatology and Organ Transplant Dept., Ciudad de Buenos Aires
- Hospital Universitario Clementino Fraga Filho, Rio de Janeiro, Brazil
- Service de Neurologie, CHU Henri Mondor, Paris, France
- Universitatsklinikum Munster, Transplant Hepatology, Münster, Germany
- Portugal (4):
  - Serviço de Neurologia-Hospital de Santa Maria, Lisbon
  - Servicio de Neurologica Piso 7, Hospital de Santa Maria, Lisbon
  - Unidade Clinica de Paramiloidose-Hospital Santo Antonio, Porto
  - Unidade Clinica de Paramiloidose, Hospital Geral de Santo Antonio, Largo Prof Abdel Salazar, Porto
- Sweden (2):
  - Umea University Hospital, Umeå
  - FAP-Teamet Familjar Amyloids, Norrlands universitetssjukhus, Umeå

REFERENCES:
- [Derived] Merlini G, Coelho T, Waddington Cruz M, Li H, Stewart M, Ebede B. Evaluation of Mortality During Long-Term Treatment with Tafamidis for Transthyretin Amyloidosis with Polyneuropathy: Clinical Trial Results up to 8.5 Years. Neurol Ther. 2020 Jun;9(1):105-115. doi: 10.1007/s40120-020-00180-w. Epub 2020 Feb 27. PMID 32107748
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- [Derived] Amass L, Li H, Gundapaneni BK, Schwartz JH, Keohane DJ. Influence of baseline neurologic severity on disease progression and the associated disease-modifying effects of tafamidis in patients with transthyretin amyloid polyneuropathy. Orphanet J Rare Dis. 2018 Dec 17;13(1):225. doi: 10.1186/s13023-018-0947-7. PMID 30558645
- [Derived] Waddington Cruz M, Amass L, Keohane D, Schwartz J, Li H, Gundapaneni B. Early intervention with tafamidis provides long-term (5.5-year) delay of neurologic progression in transthyretin hereditary amyloid polyneuropathy. Amyloid. 2016 Sep;23(3):178-183. doi: 10.1080/13506129.2016.1207163. Epub 2016 Aug 5. PMID 27494299
- [Derived] Coelho T, Maia LF, da Silva AM, Cruz MW, Plante-Bordeneuve V, Suhr OB, Conceicao I, Schmidt HH, Trigo P, Kelly JW, Labaudiniere R, Chan J, Packman J, Grogan DR. Long-term effects of tafamidis for the treatment of transthyretin familial amyloid polyneuropathy. J Neurol. 2013 Nov;260(11):2802-14. doi: 10.1007/s00415-013-7051-7. Epub 2013 Aug 22. PMID 23974642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed study FX-005 (NCT00409175), were eligible for the current study FX-006 (NCT00791492).
Groups:
- Tafamidis-Tafamidis: Participants who received tafamidis (Fx-1006A) 20 milligram (mg) capsule orally once daily for 18 months during previous study FX-005 (NCT00409175), received tafamidis (Fx-1006A) 20 mg capsule orally once daily for 12 months.
- Placebo-Tafamidis: Participants who received placebo matched to tafamidis (Fx-1006A) 20 mg capsule orally once daily for 18 months during previous study FX-005 (NCT00409175), received tafamidis (Fx-1006A) 20 mg capsule orally once daily for 12 months.
Period: Overall Study
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Started | 45 | 41
TREATED | 44 | 41
Completed | 39 | 38
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Liver transplantation | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis | Total
Number analyzed (Participants) | 44 | 41 | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13.4) | 39.6 (13.2) | 40.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment as Measured by Neuropathy Impairment Score - Lower Limb (NIS-LL) at Month 6
Description: Response to treatment indicated by either improvement(decrease from baseline) or stabilization(change from baseline of 0 to less than[<] 2) in NIS-LL score,based on mean of 2 scores in 1 week period.NIS-LL assessed muscle weakness,reflexes,sensation.Each item scored separately for left,right limbs.Components of muscle weakness:0(normal)-4(paralysis),higher score=more weakness;reflexes,sensation:0=normal,1=decreased,or 2=absent.Total NIS-LL score range 0-88,higher score=more impairment. For tafamidis-tafamidis group, NIS-LL baseline value of previous study FX-005(NCT00409175) used as reference.
Time Frame: Month 6
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study medication and had no more than 2 months interruption between studies FX-005 and FX-006. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 37 | 32
percentage of participants | 62.2 [44.8 to 77.5] | 68.8 [50.0 to 83.9]

2. Primary Outcome: Percentage of Participants With Response to Treatment as Measured by Neuropathy Impairment Score - Lower Limb (NIS-LL) at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: ITT population included all participants who received at least one dose of study medication and had no more than 2 months interruption between studies FX-005 and FX-006. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 33 | 30
percentage of participants | 54.5 [36.4 to 71.9] | 60.0 [40.6 to 77.3]

3. Primary Outcome: Change From Baseline in Norfolk Quality of Life- Diabetic Neuropathy (QOL-DN) Total Quality of Life (TQOL) Score at Month 6
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy; Item 1 to 7: related to symptoms and presence of symptoms was assessed as 1 and absence was assessed as 0. Item 8-35: related to activities of daily living and scored on a 5-point Likert scale, where 0= no problem and 4= severe problem (except item 32, where -2= much better, 0=about the same, 2=much worse). TQOL= sum of all the items, total possible score range= -2 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Month 6
Population: ITT population included all participants who received at least one dose of study medication and had no more than 2 months interruption between studies FX-005 and FX-006. 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
units on a scale
  Baseline | 21.05 (21.88) | 38.09 (31.89)
  Change at Month 6 | 0.03 (8.83) | -4.88 (15.29)

4. Primary Outcome: Change From Baseline in Norfolk Quality of Life- Diabetic Neuropathy (QOL-DN) Total Quality of Life (TQOL) Score at Month 12
Description: as for outcome 3
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 32 | 30
units on a scale | 2.25 (8.91) | -2.33 (15.66)

5. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score - Lower Limb (NIS-LL) Score at Month 6 and 12
Description: NIS-LL: assessed muscle weakness, reflexes and sensation; scored separately for left and right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) are scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) were scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS-LL score range 0-88, higher score=greater impairment.
Time Frame: Baseline, Month 6, 12
Population: ITT population included all participants who received at least one dose of study medication and had no more than 2 months interruption between studies FX-005 and FX-006. 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n' signifies participants for this measure at specified time point for each arm group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
units on a scale
  Baseline (n=38,33) | 8.38 (13.23) | 17.50 (20.82)
  Change at Month 6 (n=37,32) | 0.93 (3.65) | 1.89 (4.55)
  Change at Month 12 (n=33,30) | 1.36 (4.77) | 1.60 (8.20)

6. Secondary Outcome: Change From Baseline in Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Domain Scores at Month 6 and 12
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire to assess impact of DN on QOL; Item 1-7:scored as 1=symptoms present, 0=symptoms absent. Item 8-35:scored on 5-point Likert scale: 0=no problem,4=severe problem (except item 32: -2=much better, 0=about same, 2=much worse). Norfolk QOL-DN summarized in 5 domains(score range):physical functioning/large fiber neuropathy(-2 to 58), activities of daily living(ADLs) (0 to 20), symptoms(0 to 32), small fiber neuropathy(0 to 16), autonomic neuropathy(0 to 12); higher score=greater impairment,for each. Total score=-2 to138(higher score=worse QOL).
Time Frame: Baseline, Month 6, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
units on a scale
  Baseline: physical functioning (n=38,33) | 9.45 (11.43) | 19.88 (17.44)
  Baseline: ADLs (n=38,33) | 2.21 (4.38) | 3.48 (5.13)
  Baseline: symptoms (n=38,33) | 5.34 (4.43) | 7.48 (5.48)
  Baseline: small fiber neuropathy (n=38,33) | 2.50 (3.85) | 4.42 (4.23)
  Baseline: autonomic neuropathy (n=38,33) | 1.55 (2.37) | 2.82 (3.12)
  Change at Month 6: physical functioning (n=37,32) | 0.14 (4.08) | -3.00 (8.08)
  Change at Month 6: ADLs (n=37,32) | -0.30 (1.45) | -0.59 (3.02)
  Change at Month 6: symptoms (n=34,32) | 0.00 (3.18) | -0.75 (4.27)
  Change at Month 6: small fiber neuropathy(n=37,32) | -0.14 (2.64) | -0.09 (2.32)
  Change at Month 6: autonomic neuropathy (n=37,32) | 0.19 (1.33) | -0.44 (2.00)
  Change at Month 12: physical functioning(n=32,30) | 1.84 (6.00) | -0.83 (9.62)
  Change at Month 12: ADLs (n=32,30) | 0.13 (1.01) | -0.50 (3.35)
  Change at Month 12: symptoms (n=32,30) | -0.66 (2.54) | -1.10 (3.32)
  Change at Month 12:small fiber neuropathy(n=32,30) | 0.41 (2.87) | 0.40 (2.61)
  Change at Month 12: autonomic neuropathy (n=32,30) | 0.53 (1.46) | -0.30 (1.66)

7. Secondary Outcome: Change From Baseline in Summated 7 Score for Large Nerve Fiber Function at Month 6 and 12
Description: Summated 7 score: composite score included five Nerve Conduction Studies (NCS) attributes (peroneal nerve distal motor latency, peroneal nerve compound muscle action potential, peroneal nerve motor conduction velocity, tibial nerve distal motor latency, and sural nerve sensory nerve action potential amplitude) along with Vibration Detection Threshold (VDT) obtained in great toes, and Heart Rate Response to Deep Breathing (HRDB) value. Score was determined through reference to normal values for age, sex and height. Total score range= -26 to 26, where higher score=worse nerve function.
Time Frame: Baseline, Month 6, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
units on a scale
  Baseline (n=38,33) | 6.68 (8.51) | 10.06 (10.68)
  Change at Month 6 (n=37,32) | -0.01 (2.99) | 1.38 (3.58)
  Change at Month 12 (n=33,30) | 0.64 (3.23) | 1.48 (4.02)

8. Secondary Outcome: Change From Baseline in Summated 3 Score for Small Nerve Fiber Function at Month 6 and 12
Description: Summated 3 Nerve Tests Small Fiber Normal Deviates Score (NTSFnds) included cooling threshold for the lower limbs, heat pain threshold for the lower limbs and HRDB. Total score range= -11.2 to 11.2, where higher score=worse nerve function.
Time Frame: Baseline, Month 6, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
units on a scale
  Baseline (n=38,33) | 4.78 (4.33) | 7.08 (4.39)
  Change at Month 6 (n=36,32) | 0.43 (1.51) | 0.38 (1.08)
  Change at Month 12 (n=32,30) | 0.59 (1.28) | 0.50 (1.48)

9. Secondary Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Month 6 and 12
Description: BMI was calculated by weight divided by height squared. mBMI was calculated by multiplying BMI by serum albumin levels to compensate for edema formation. A progressive decline in mBMI indicated worsening of disease severity.
Time Frame: Baseline, Month 6, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: (kilogram/square meter)*(gram/liter)
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 33
(kilogram/square meter)*(gram/liter)
  Baseline (n=38,33) | 23.94 (2.97) | 22.71 (5.15)
  Change at Month 6 (n=37,32) | -0.13 (0.81) | 0.42 (1.14)
  Change at Month 12 (n=33,30) | -0.12 (1.16) | 0.73 (1.45)

10. Secondary Outcome: Change From Baseline in Troponin I Concentration at Week 6, Month 3, 6 and 12
Description: Troponin I was biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ left ventricular [LV] wall stress).
Time Frame: Baseline, Week 6, Month 3, 6, 12
Population: Safety population included participants who received at least one dose of study medication. 'N' (number of participants analyzed) signifies participants evaluable for this measure. 'n' signifies participants evaluable for this measure at the specified time point for each arm group.
Measure: Median (Full Range); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 29 | 30
nanogram/milliliter (ng/mL)
  Baseline (n=29,30) | 0.2 [0.2 to 0.5] | 0.2 [0.2 to 0.2]
  Change at Week 6 (n=28,29) | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.0]
  Change at Month 3 (n=29,30) | 0.0 [-0.1 to 0.3] | 0.0 [0.0 to 0.7]
  Change at Month 6 (n=29,30) | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 0.1]
  Change at Month 12 (n=26,28) | 0.0 [-0.3 to 0.4] | 0.0 [0.0 to 0.0]

11. Secondary Outcome: Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration at Week 6, Month 3, 6 and 12
Description: NT-proBNP was biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ LV wall stress).
Time Frame: Baseline, Week 6, Month 3, 6, 12
Population: as for outcome 10
Measure: Median (Full Range); unit: picogram/milliliter (pg/mL)
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 33 | 34
picogram/milliliter (pg/mL)
  Baseline (n=33,34) | 41.0 [19.0 to 2879.0] | 75.0 [20.0 to 1127.0]
  Change at Week 6 (n=33,33) | 6.0 [-650.0 to 525.0] | -1.0 [-292.0 to 97.0]
  Change at Month 3 (n=33,34) | 11.0 [-52.0 to 1355.0] | 1.0 [-514.0 to 229.0]
  Change at Month 6 (n=33,33) | 9.0 [-210.0 to 3878.0] | 0.0 [-473.0 to 170.0]
  Change at Month 12 (n=30,29) | 15.0 [-104.0 to 3840.0] | -6.0 [-342.0 to 410.0]

12. Secondary Outcome: Intraepidermal Nerve Fiber (IENF) Density
Description: IENF density was quantified in 3 millimeter (mm) immunostained skin punch biopsies containing epidermis and superficial dermis to evaluate the amount and morphological appearance of small diameter nerve fibers, both somatic and autonomic, in sensory neuropathies. It is used in diagnosing various neuropathic conditions.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 11 | 5
fibers/mm
  Left distal leg | 8.2 (9.8) | 8.0 (9.2)
  Left proximal thigh | 16.1 (12.6) | 15.3 (11.9)

13. Secondary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR) Tetramer
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The Fraction of Initial (FOI) is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI.
Time Frame: Month 6, 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 36 | 32
percentage of participants
  Month 6 | 94 [81 to 99] | 97 [83 to 99]
  Month 12 | 94 [80 to 99] | 93 [77 to 99]

14. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE: AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent/significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug, up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after last dose of study medication
Population: Safety population included participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 44 | 41
participants | 5 | 4

15. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events Greater Than or Equal to Grade 3
Description: AE=any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 (Death) events=death related to an AE. Treatment-emergent events=between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after last dose of study medication
Population: Safety population included participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 44 | 41
participants | 6 | 4

16. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-emergent Echocardiography (ECHO) Findings
Description: Clinically significant ECHO findings included: LV posterior wall thickness greater than or equal to (>=)13 mm, LV septal thickness >= 13 mm, right ventricular thickness >= 7 mm, ratio of peak mitral early diastolic and atrial contraction velocity (E/A ratio) >= 2, prime septal (E/E) >15, ejection fraction < 50 percent (%), E deceleration time <= 150 millisecond (ms), isovolumic relaxation time (IVRT) <= 70 ms, any valve thickening (> trace regurgitation in mitral, aortic, pulmonary, or tricuspid valves), abnormal respiratory variation of inferior vena cava, pericardial effusion.
Time Frame: Baseline, Day 1 up to Month 12 (anytime on-treatment)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 38 | 34
participants
  Baseline (n=38,34) | 23 | 18
  Anytime on-treatment (n=21,23) | 16 | 13

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings
Description: Clinically significant ECG findings included: corrected QT (QTc) > 450 ms, QTc >500 ms, change in QTc between 30 and 60 ms, change in QTc greater than or equal to 60 ms.
Time Frame: Baseline, Day 1 up to Month 12 (anytime on-treatment)
Population: Safety population included participants who received at least one dose of study medication. 'n' signifies participants for this measure at specified time point for each arm group.
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 44 | 41
participants
  Baseline (n=44,41) | 16 | 17
  Anytime on-treatment (n=28,24) | 6 | 6

18. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-emergent Holter Monitor Findings
Description: Clinically significant Holter monitor findings included: atrial fibrillation/flutter, atrial tachycardia, non-sustained ventricular tachycardia (<30 beats), sustained ventricular tachycardia (>= 30 beats), sinus pause (RR >2.0 second, where RR=60/heart rate), ventricular premature contractions.
Time Frame: Baseline, Day 1 up to Month 12 (anytime on-treatment)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 44 | 41
participants
  Baseline (n=44,41) | 20 | 21
  Anytime on-treatment (n=24,20) | 8 | 7

19. Other Pre Specified Outcome: Number of Participants Who Discontinued Due to Clinical or Laboratory Adverse Events
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 12
Population: Safety population included participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Number analyzed (Participants) | 44 | 41
participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tafamidis-Tafamidis | Placebo-Tafamidis
Serious Adverse Events (participants affected / at risk) | 5/44 | 4/41
Other Adverse Events (participants affected / at risk) | 24/44 | 24/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis-Tafamidis (N=44) | Placebo-Tafamidis (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Blood electrolytes decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis-Tafamidis (N=44) | Placebo-Tafamidis (N=41)
Punctate keratitis (Eye disorders) | 3 | 3
Dry eye (Eye disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 2 | 4
Urinary tract infection (Infections and infestations) | 5 | 6
Influenza (Infections and infestations) | 3 | 7
Nasopharyngitis (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Thermal burn (Injury, poisoning and procedural complications) | 4 | 4
Headache (Nervous system disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 1 | 5

LIMITATIONS AND CAVEATS:
Instead of intended endpoint 'heat pain and cooling threshold', results of 'summated 3 score for small nerve fiber function' were reported. Designation of outcomes as primary and secondary was based on study team input as study did not specify this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.